Effect of exercise in obese patients with chronic kidney diseases

NCT number: P.T. REC/012/002608.

Date: 1/5/2020

**Statistical analysis:** 

Pre and post treatment measures analyzed by Minitab version 18 (LLC headquartered in state

college Pennsylvania, USA). All the data presented as the mean ±SD. An independent t-test was

used to compare between the variables of the participants. Paired t-test was used to compare

between pretreatment and post treatment values of the physical performance and obesity of both

groups, and independent t- test was used to compare between both groups. The significance level

was set at  $P \le 0.05$  for all tests.

**Results:** 

60 patients 26 male (43.3%) and 34 female (56.7%). Age between 35 and 60. There is no significant

difference between both groups in age P= 0.708. Also no significant difference in BMI in both

groups 33.8 and 33.96, WC 141.67 and 146.26. WHR0.91 and 0.92, TUG24.46 and 28.3, STS5

32.7 and 31.8, STS60, 9.13 and 8.13, 6MWD,246.13 and 215.17, systolic blood pressure 156.3 and

160.5, diastolic blood pressure 85.8 and 84.7, mean blood pressure 115.3 and 118.8, heart rate 76

and 76.3, blood glucose 197.7 and 189.47.

After three months of exercises BMI in both groups 31.7 and 31.8, WC 130.57 and 137.33. WHR

0.85 and 0.88, TUG18.4 and 21.3, STS5 20.9 and 19.5, STS60, 14.6 and 14.2, 6MWD, 343.5 and

338.5, systolic blood pressure 133.8 and 132.0, diastolic blood pressure 75.5 and 72.7, mean blood

pressure 92.4 and 105.8, heart rate 76 and 76.3, blood glucose 178.6 and 183.6.

Table (1): pre and post measurements of group1

| Item | Pretreatment group 1 Post treatment group 1 | | T test | P value |
|---|---|---|---|---|
| | | | 1 test | |
| BMI (kg//m <sup>2</sup> ) | 33.8±1.99 | 31.7± 2.88 | 2.72 | 0.011 |
| Waist circumference(WC) (cm) | 141.67±16.39 | 130.57± 10.22 | 3.90 | 0.001 |
| Waist to hip(WHR) | 0.91367±0.03409 | 0.85633± 0.04522 | 15.58 | 0.000 |
| Time up and go(TUG) (sec) | 24.46±4.023 | 18.4±2.40 | 9.51 | 0.000 |
| Sit to stand test(STS5) (sec) | 32.067±3.562 | 20.867± 3.014 | 23.67 | 0.000 |
| STS60 (cycle/min) | 9.133±1.167 | 14.567± 2.096 | -15.05 | 0.000 |
| 6minutes walk distance (6MWD) | 246.13±17.48 | 343.50± 22.25 | -19.78 | 0.000 |
| (m) | | | | |
| Systolic blood pressure(mm Hg) | 156.33±7.76 | 133.83 ± 5.83 13.8 | | 0.000 |
| Diastolic blood pressure (mm Hg) | 85.833±4.170 | 75.500± 4.798 | 16.37 | 0.000 |
| Mean blood pressure (mm Hg) | 115.33±7.60 | 92.40±4.60 | 16.43 | 0.000 |
| Heart rate(beat/min) | 76.000±2.213 | 71.567± 1.478 | 11.41 | 0.000 |
| Blood glucose (mg/dl) | 197.7±3.49 | 178.57±7.00 | 11.28 | 0.000 |

Table (2) pre and post measurements of group2

| Table (2) pre and post measuremen | its of groups | | | |
|---|---|---|---|---|
| Item | m Pretreatment Post treatment group 1 group 1 | | T test | P value |
| BMI (kg//m <sup>2</sup> ) | 33.96±2.55 | 31.86±2.98 | 3.58 | 0.001 |
| Waist circumference(WC) (cm) | 146.27±9.58 | 137.33±10.74 | 8.36 | 0.000 |
| Waist to hip(WHR) | 0.92600±0.03450 | 0.88667±0.03633 | 15.52 | 0.000 |
| Time up and go(TUG) (sec) | 28.3±1.985 | 21.267±2.434 | 15.42 | 0.000 |
| Sit to stand test(STS5) (sec) | 31.800±5.346 | 19.533±4.158 | 17.45 | 0.000 |
| STS60 (cycle/min) | 8.133±1.137 | 14.167±1.704 | -21.43 | 0.000 |
| 6minutes walk distance (6MWD) | 215.17±54.36 | 338.53±26.22 | -10.00 | 0.000 |
| (m) | | | | |
| Systolic blood pressure(mm Hg) | 160.50±8.34 | 132.00±6.38 | 15.33 | 0.000 |
| Diastolic blood pressure (mm Hg) | 84.667±4.138 | 72.667±4.097 | 15.37 | 0.000 |
| Mean blood pressure (mm Hg) | 118.77±6.70 | 105.83±21.16 | 3.49 | 0.002 |
| Heart rate(beat/min) | 76.300±1.725 | 70.367±0.615 | 19.34 | 0.000 |
| Blood glucose (mg/dl) | 198.47±1.98 | 183.63±4.71 | 16.37 | 0.000 |

Table (3) post measurements of both groups

| Item | Pretreatment group 1 | Post treatment group 1 | T test | P value |
|---|---|---|---|---|
| BMI (kg//m <sup>2</sup> ) | 31.733±2.888 | 31.867±2.980 | -0.15 | 0.881 |
| Waist circumference(WC) (cm) | 130.57±10.22 | 137.33±10.74 | -2.78 | 0.009 |
| Waist to hip(WHR) | 0.85633±0.04522 | 0.88667±0.03633 | -2.87 | 0.008 |
| Time up and go(TUG) (sec) | 18.400±2.401 | 21.267±2.434 | -5.11 | 0.000 |

| Sit to stand test(STS5) (sec) | 20.867±3.014 | 19.533±4.158 | 1.20 | 0.240 |
|---|---|---|---|---|
| STS60 (cycle/min) | 14.567±2.096 | 14.167±1.704 | 0.89 | 0.380 |
| 6minutes walk distance (6MWD) | 343.50±22.25 | 338.53±26.22 | 0.80 | 0.433 |
| (m) | | | | |
| Systolic blood pressure(mm Hg) | 133.83±5.83 | 132.00± 6.38 | 1.07 | 0.295 |
| Diastolic blood pressure (mm Hg) | 75.500±4.798 | 72.667±4.097 | 2.25 | 0.032 |
| Mean blood pressure (mmHg) | 92.40±4.60 | 105.83±21.16 | -3.21 | 0.003 |
| Heart rate(beat/min) | 71.567±1.478 | 70.367±0.615 | 4.09 | 0.000 |
| Blood glucose (mg/dl) | 178.57±7.00 | 183.63±4.71 | 3.18 | 0.003 |